CLINICAL TRIAL: NCT00260312
Title: Randomized Placebo-Controlled Trial of Inactivated Poliovirus Vaccine in Cuba
Brief Title: Study of Inactivated Poliovirus Vaccine Given at an Earlier Schedule With Shorter Intervals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pan American Health Organization (Other)
Collaborators: World Health Organization (Other); Institute Pedro Kouri, Ministry of Public Health (Cuba) (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3827
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2004-01

CONDITIONS: Level of Immunity Against Poliovirus Infection
Keywords: inactived; polio; vaccine; cuba; trial; randomized; eradication
MeSH Terms: conditions — Poliomyelitis

INTERVENTIONS:
Biological: Inactivated Polio Vaccine given at an accelerated schedule

SUMMARY:
The purpose of this study was to evaluated the effectiveness of inactivated poliovirus vaccine at a vaccine schedule that is commonly used in developing countries. The effectiveness of inactivated poliovaccine given at this schedule is important to national policy makers as they consider vaccination policies after the use of oral polio vaccine is discontinued.

DETAILED DESCRIPTION:
After polio eradication, access to live polioviruses will be highly restricted, and oral poliovirus vaccine (OPV) use must be discontinued. OPV-using countries must decide whether to switch to inactivated poliovirus vaccine (IPV) or stop polio vaccination. Because only limited data are available on IPV immunogenicity in tropical developing countries, we conducted a randomized controlled trial of IPV in Cuba. The objectives of this study were to assess the humoral and mucosal immunogenicity conferred by IPV administered at the WHO-EPI schedule (6,10,14 wks of age) vs. placebo. A third arm was added to evaluate the immunogenicity of IPV administered at 2 and 4 months of age. Antibody titers were measured prior to the first dose as well as 1 month after the last dose in each study arm. Target sample size was 100 children in each arm. Mucosal (intestinal immunity) was measured indirectly through assessing poliovirus excretion in each group after a "natural challenge" of trivalent oral polio vaccine (OPV)recieved by study participants through their participation in the annual OPV mass campaigns approximately 1 month after their last dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

Infants born 18 - 20 weeks prior to the first round of the 2002 National Immunization Days in cuba (in March 2002).

Born healthy at one of the 4 designated maternity hospitals in Cuba

Exclusion Criteria:

Serious congenital defect/disease at birth

-

Ages: 6 Weeks to 2 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Start 2001-08; Study Completion 2003-01

PRIMARY OUTCOMES:
Seroconversion by measuring level of poliovirus antibodies in serum. Also, measure of virus titer in stools to indirectly assess the level of intestinal mucosal immunity

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Galindo, MD, Principal Investigator — Ministry of Public Health, Cuba

REFERENCES:
- [Derived] Cuba IPV Study Collaborative Group. Randomized, placebo-controlled trial of inactivated poliovirus vaccine in Cuba. N Engl J Med. 2007 Apr 12;356(15):1536-44. doi: 10.1056/NEJMoa054960. PMID 17429085